CLINICAL TRIAL: NCT05250453
Title: Cardiopulmonary Resuscitation; Epidemiology, Quality, Survival and Injuries.
Brief Title: Quality of the Cardio-pulmonary Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: National Istitute For Health and Welfare, Finland (Other Government)
Responsible Party: Sponsor
Other Study IDs: R18100; R18163 (Registry Identifier: ResusciCPC); R21124 (Registry Identifier: ResusciCT)
Record Dates: First submitted 2022-01-03; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: CPR, injuries, OHCA
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cardiac arrest: All patients having sudden cardiac arrest out-of-hospital in Pirkanmaa, Finland
- ResusInj: OHCA survivors having CPR related injuries or carotid stenosis analyzed by CT
- ResusCPC: OHCA survivors neurological outcome

SUMMARY:
Patients having sudden cardiac arrest have very poor prognosis. It is devastating for patient and family. But also very expensive for nations economics when working-age people die or disable due to cardiac arrest. Recent studies have shown that high quality of cardiopulmonary resuscitation (CPR) and minimized delays increases the survival after cardiac arrest. In this objective prospective study we will use Zoll´s X Series defibrillator on every emergency medicine systems (EMS´s) unit in Pirkanmaa area, Finland, to collect information on CPR quality. Real CPR Help® will collect the information on depth, frequency and pauses during CPR. We will make an Utstein analysis on OHCA during one year period and compare the results on Utstein analysis made in the same area on 2013-2014. We will analyse the quality of CPR and compare it to the outcome from OHCA and neurological outcome 3 months after resuscitation. In addition we will analyse the CPR related injuries and compare these to the compression depth and number of persons performing CPR.

In one part of the study we will evaluate the incidence of OHCA in different risk areas of Pirkanmaa and analyse the influence of time delay and location to the outcome out of hospital and neurological outcome 3 months after resuscitation. We will also analyse if the time of post-resuscitation care before getting to the hospital or stenosis in carotid artery affects the outcome from OHCA and neurological outcome 3 months after resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest
* > 18 years of age

Exclusion Criteria:

* < 18 years of age
* prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cardiac arrest patients in Etelä-Pohjanmaa and Pirkanmaa, Finland
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
QualityCPR | 1 year
  The success rate of current guidelines (depth and frequency of chest compression, epidemiology)
Neurological survival after CA | 3 months after OHCA
  Neurological survival after CA

SECONDARY OUTCOMES:
CPR related injuries | 1 year
  Injuries detected in CT scanning or in autopsy
Stenosis of the carotid artery | 3 months after OHCA
  Effect of the carotid artery stenosis to the neurological survival. Survivals having CPC 1-2 prior to the cardiac arrest and are taken to the ICU are scanned with carotid CTA after informed consent. The degree of stenosis will be compared to the CPC-level 3monts aften OHCA.
the dispatch calls concerning OHCA | 1 year
  Analyze the key words and dispatch assisted CPR through the emergency call. All emergency call conserning OHCA patients will be listened. We will analyze the keywords which are used by layperson to describe patient having cardiac arrest.
  We will also analyze the amount of given dispatch assisted CPR and compare the amount to the primary rythm.
the quality of the postresuscitation care | 3 months after OHCA
  The correlation of the duration and the quality of the postresuscitation care before getting in to the hospital and the outcome from OHCA

CONTACTS AND LOCATIONS:
Overall Officials: Piritta Setälä, PhD, Study Director — Tampere University Hospital; Sanna Hoppu, PhD, Study Director — Tampere University Hospital; Jyrki Ollikainen, MD, Principal Investigator — Tampere University Hospital; Kati Järvelä, PhD, Study Director — Tampere University Hospital; Valtteri Järvenpää, MB, Principal Investigator — Tampere University Hospital; Ville Jalkanen, PhD, Study Director — Tampere University Hospital; Joonas Tirkkonen, PhD, Study Director — Tampere University Hospital; Heini Huhtala, PhD, Study Director — Tampere University; Mika Martiskainen, PhD, Study Director — Finnish Institute for Health and Welfare; Riikka Nevalainen, MD, Study Director — Tampere University Hospital
Locations (1):
- Tampere University hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No